CLINICAL TRIAL: NCT01576848
Title: Impact of Carbohydrate Co-ingestion on the Post-prandial Anabolic Response of Protein in Young and Elderly Men
Acronym: PRO-CARB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Henrike Hamer, MSc, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: METC 11-3-040
Record Dates: First submitted 2011-08-09; First posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Sarcopenia
Keywords: muscle metabolism; intrinsically labeled protein; protein synthesis; insulin; perfusion
MeSH Terms: conditions — Sarcopenia; Insulin Resistance | interventions — Proteins; Carbohydrates; Caseins; Glucose; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GROUP 1 (OLD-PRO) (Experimental): test drink contains intrinsically labeled protein alone
  Interventions: Dietary Supplement: Protein
- GROUP 2 (OLD-PRO/CARB) (Experimental): test drink contains intrinsically labeled protein and carbohydrate
  Interventions: Dietary Supplement: Protein + carbohydrate
- GROUP 3 (YOUNG-PRO) (Experimental): test drink contains intrinsically labeled protein alone
  Interventions: Dietary Supplement: Protein
- GROUP 4 (YOUNG-PRO/CARB) (Experimental): test drink contains intrinsically labeled protein and carbohydrate
  Interventions: Dietary Supplement: Protein + carbohydrate

INTERVENTIONS:
Dietary Supplement: Protein — Subjects will receive a drink containing 20 gram intrinsically labelled casein.
  Half of the subject are young males (YOUNG)(age between 18 and 35 y) and half of the subjects are elderly males (OLD)(age between 70 and 85 y).
  Other Names: Intrinsically labelled casein
  Arms: GROUP 1 (OLD-PRO); GROUP 3 (YOUNG-PRO)
Dietary Supplement: Protein + carbohydrate — subjects will receive a drink containing 20 gram intrinsically labelled casein plus 60 gram carbohydrates.
  Half of the subject are young males (YOUNG)(age between 18 and 35 y) and half of the subjects are elderly males (OLD)(age between 70 and 85 y).
  Other Names: Casein plus dextrose monohydrate and maltodextrin
  Arms: GROUP 2 (OLD-PRO/CARB); GROUP 4 (YOUNG-PRO/CARB)

SUMMARY:
Rationale: Age related muscle loss (sarcopenia) is assumed to be related to the impaired postprandial muscle protein synthetic response to protein and/or amino acid administration in the elderly vs the young. Co-ingestion of carbohydrate increases post-prandial insulin secretion. Insulin affects skeletal muscle blood flow and may therefore affect substrate availability and postprandial muscle protein synthesis. However, it is unclear whether the response to the combined intake of protein and carbohydrates is different in elderly compared to young subjects.

Hypothesis: Adding carbohydrate to a bolus of protein represents an effective strategy to overcome the impaired postprandial muscle protein synthesis in the elderly.

Objective: The primary objective of the study is to investigate whether carbohydrate co-ingestion augments the in vivo postprandial muscle protein synthetic response after protein ingestion and whether this response is different between young and elderly subjects. The secondary objective of the study is to assess the effect of carbohydrate co-ingestion on insulin levels and microvascular perfusion in young and elderly subjects.

Intervention: The intervention consists of a single test day during which the subjects will receive a drink containing 20 gram intrinsically labelled casein with or without 60 gram carbohydrates. In addition, continuous intravenous tracer infusions of labeled amino acids will be administered. During the test day 18 plasma samples and 4 muscle biopsies will be collected over a period of 8½ h. Furthermore, muscle skeletal blood flow will be estimated using sidestream darkfield imaging (SDF) in sublingual position.

DETAILED DESCRIPTION:
With human aging, there is a gradual but progressive decline in skeletal muscle tissue, also known as sarcopenia . Sarcopenia is accompanied by a reduced physical performance, the loss of functional capacity, increased risk of falling and increased likelihood of developing chronic metabolic diseases, such as type 2 diabetes and obesity. Eventually this also results in increased hospitalisation and institutionalization of elderly in nursing homes, and high health care costs. Therefore, it is important to investigate approaches to diminish the loss of skeletal muscle mass during aging. To preserve muscle mass, protein intake is important, because it provides the building blocks for muscle tissue: amino acids. Since basal muscle protein synthesis rates do not seem to differ between young and elderly, currently many research groups focus on postprandial muscle protein synthesis. Skeletal muscle protein synthesis has been shown to be highly dependent on protein intake. However, recent data indicate that the muscle protein synthetic response to protein intake is attenuated in the elderly. A blunted postprandial muscle protein synthetic response over a prolonged period might result in diminished muscle protein accretion and could eventually contribute to sarcopenia.

The anabolic response to protein intake appears to be mainly mediated by an elevation of plasma essential amino acids. In addition, ingestion of carbohydrate leads to an attenuation of muscle protein breakdown by virtue of an elevation in plasma insulin, further promoting positive net protein balance. This is mediated by insulin's known action of increasing muscle blood flow and thereby augmenting muscle substrate delivery, which may lead to further stimulation of muscle protein synthesis. It has been shown that there is an insulin resistance with respect to muscle protein anabolism in elderly compared to young subjects during conditions of high plasma amino acid and insulin availability. This suggests that the reduced ability of insulin to augment muscle microvascular perfusion decreases the amino acid stimulus.

In the present study the investigators will assess the effect of a single meal-like amount of intact protein with or without carbohydrates on post-prandial muscle protein synthesis in the elderly (70-85 y) compared to the young (18 - 30 y). Furthermore, the investigators are going to investigate whether the muscle protein synthetic response is associated with an increase in the microvascular perfusion after ingestion of the meal using Sidestream Dark Field (SDF) imaging. SDF measurements will be taken in de oral cavity underneath the tongue, since this area is easily accessible and is representative for microvascular perfusion. To be able to measure the effect of protein ingestion on muscle protein synthesis the investigators will use intrinsically labelled casein. This allows us to determine the true incorporation of amino acids from the ingested, intact casein into the muscle, taken into account the influence of digestion and absorption processes of a whole protein. Intrinsically labelled milk proteins were derived from milk that has been collected from cows that were infused with L-[1-13C] phenylalanine.

The following hypotheses will be investigated:

1. The combined intake of protein and carbohydrates augments post-prandial muscle protein synthesis in the elderly, but not in the young subjects.
2. The increased insulin production following the combined intake of protein and carbohydrates results in an increased microvascular perfusion that is related to the post-prandial muscle protein synthetic response.

ELIGIBILITY:
Inclusion criteria:

* Males
* Age 70-85 years or Age 18-30 years
* BMI < 30 kg∙m2

Exclusion criteria:

* Diabetes
* HbA1c > 7.0%
* Obesity (BMI > 30 kg/m2)
* Diagnosed impaired renal or liver function
* All co-morbidities interacting with mobility and muscle metabolism of the lower limbs (e.g. arthrosis, arthritis, spasticity/rigidity, all neurological disorders and paralysis).
* Hypertension (according to WHO criteria) (36)
* Use of anticoagulants, blood diseases, allergy for lidocain
* Use of NSAIDs and acetylsalicylic acid
* Use of gastric acid inhibitors
* Patients suffering from PKU (Phenylketonuria)
* Participation in any regular exercise program
* Unstable body weight over the last 3 months

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change from fasted state in Muscle protein synthesis rate (expressed as Fractional Synthetic Rate, FSR) at different time points postprandial | Participants will be followed in a fasted state over 2 hours and in a postprandial state over 5 hours

SECONDARY OUTCOMES:
Change from fasted state in Whole body protein balance at different time ponits postprandial | Participants will be followed in a fasted state over 2 hours and in a postprandial state over 5 hours
Change from fasted state in Microvascular perfusion at different time points postprandial | Participants will be followed in a fasted state over 2 hours and in a postprandial state over 5 hours
Change from fasted state in Digestion kinetics of dietary intrinsically labeled protein at different time points postprandial | Participants will be followed in a fasted state over 2 hours and in a postprandial state over 5 hours
Change from fasted state in Absorption kinetics of dietary intrinsically labeled protein at different time points postprandial | Participants will be followed in a fasted state over 2 hours and in a postprandial state over 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, Prof., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Gorissen SHM, Trommelen J, Kouw IWK, Holwerda AM, Pennings B, Groen BBL, Wall BT, Churchward-Venne TA, Horstman AMH, Koopman R, Burd NA, Fuchs CJ, Dirks ML, Res PT, Senden JMG, Steijns JMJM, de Groot LCPGM, Verdijk LB, van Loon LJC. Protein Type, Protein Dose, and Age Modulate Dietary Protein Digestion and Phenylalanine Absorption Kinetics and Plasma Phenylalanine Availability in Humans. J Nutr. 2020 Aug 1;150(8):2041-2050. doi: 10.1093/jn/nxaa024. PMID 32069356
- [Derived] Kouw IW, Gorissen SH, Burd NA, Cermak NM, Gijsen AP, van Kranenburg J, van Loon LJ. Postprandial Protein Handling Is Not Impaired in Type 2 Diabetes Patients When Compared With Normoglycemic Controls. J Clin Endocrinol Metab. 2015 Aug;100(8):3103-11. doi: 10.1210/jc.2015-1234. Epub 2015 Jun 2. PMID 26037513
- [Derived] Gorissen SH, Burd NA, Hamer HM, Gijsen AP, Groen BB, van Loon LJ. Carbohydrate coingestion delays dietary protein digestion and absorption but does not modulate postprandial muscle protein accretion. J Clin Endocrinol Metab. 2014 Jun;99(6):2250-8. doi: 10.1210/jc.2013-3970. Epub 2014 Mar 14. PMID 24628553